CLINICAL TRIAL: NCT01104454
Title: Placenta and Cord Blood Analyses
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 111576
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: healthy pregnant women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — placenta, umbilical cord and cord blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to standardize methods in collecting and processing placenta, umbilical cord and cord blood samples. Samples will be used to determine potential differences between normal weight, overweight and obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* at least 7 months pregnant
* 18 years of age or older

Exclusion Criteria:

* underweight (BMI<18.5)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are at least 7 months pregnant
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Placenta, cord blood and umbilical analyses | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Saben J, Zhong Y, Gomez-Acevedo H, Thakali KM, Borengasser SJ, Andres A, Shankar K. Early growth response protein-1 mediates lipotoxicity-associated placental inflammation: role in maternal obesity. Am J Physiol Endocrinol Metab. 2013 Jul 1;305(1):E1-14. doi: 10.1152/ajpendo.00076.2013. Epub 2013 Apr 30. PMID 23632636